CLINICAL TRIAL: NCT04751747
Title: The Role of Adaptive Radiation Planning in Patients With Non-Small Cell Lung Cancer on Radiation Induced Toxicity
Brief Title: Adaptive Radiation Planning for the Reduction of Radiation-Induced Toxicity in Patients With Stage II-IV Non-small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Salma Jabbour, MD, Professor, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro2020002153; NCI-2020-08292 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2020002153; 032009 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2020-12-23; First posted 2021-02-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Lung Non-Small Cell Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Unresectable Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (CT simulation, contrast agent) (Experimental): Patients undergo CT stimulation with or without IV contrast over 1.5 hours on days -15 to -1, then undergo SOC chemoradiation on days 1-40. Patients also undergo additional CT scan simulations without IV contrast over 20 minutes each on days 15 and 29.
  Interventions: Procedure: Computed Tomography; Other: Contrast Agent

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT simulation
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Contrast Agent — Given IV
  Other Names: Contrast; Contrast Drugs; contrast material; Contrast Medium

SUMMARY:
This phase II trial studies the effect of adaptive radiation planning in reducing side effects associated with radiation treatment and immunotherapy in patients with stage II-IV non-small cell lung cancer. Prior to radiation, patients undergo simulation, where they are positioned on the treatment table in a manner that can be reproduced each time they receive treatment in order to reach the tumor exactly at the same spot each time. However, a patient's tumor may shrink as they receive radiation, exposing healthy tissue to radiation as well. Adaptive radiation planning involves re-designing a treatment plan at set intervals. The purpose of this study is to see whether establishing set time points through adaptive radiation planning, regardless of whether the doctor notices a significant decrease in tumor size, will reduce some of the side effects associated with radiation treatment and immunotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether implementing set intervals for radiation replanning reduces cardiopulmonary toxicity and preserves healthy lung and heart tissue, with the intention of establishing a new standard treatment modality.

OUTLINE:

Patients undergo computed tomography (CT) stimulation with or without intravenous (IV) contrast over 1.5 hours on days -15 to -1, then undergo standard of care (SOC) chemoradiation on days 1-40. Patients also undergo additional CT scan simulations without IV contrast over 20 minutes each on days 15 and 29.

After completion of study, patients are followed up at 3-12 weeks, and then every 6 months for approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information
* Histologically or cytological evidence of locally advanced, biopsy-proven, stage II (inoperable), III-or oligometastatic stage IV NSCLC planned to be treated with chemoradiation with concurrent or adjuvant immunotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ and marrow laboratory values for radiation therapy deemed by appropriate the investigator obtained within 14 days prior to registration for protocol therapy
* Women of childbearing potential (WOCBP) must obtain a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) at day -30 to day 0
* Women of childbearing potential must be willing to abstain from heterosexual activity or use an effective method of contraception during the time of the study period
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year

Exclusion Criteria:

* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the site investigator
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial
* Active central nervous system (CNS) metastases (if symptomatic or without prior brain imaging, subjects must undergo a head computed tomography [CT] scan or brain magnetic resonance imaging [MRI] within 28 days prior to registration for protocol therapy to exclude brain metastases)
* Treatment with any investigational agent within 28 days prior to registration for protocol therapy
* Prior chemotherapy, adjuvant therapy, or radiotherapy for lung cancer other than standard concurrent chemoradiation or up to 2 cycles of consolidation therapy
* Active second cancers
* History of psychiatric illness or social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Determine if adaptive radiation therapy reduces radiation induced pneumonitis rates | At 6 months post chemoradiation
  Will be analyzed using a one-sided z-test to determine if reduction in radiation doses to organs at risk compared will result in a lower rate of pneumonitis compared to historical controls.

SECONDARY OUTCOMES:
Determine if adaptive radiation therapy reduces radiation doses to heart and lung | Baseline up to day 29 of treatment
  Will be compared to computed tomography simulation without adaptation of lung tumor volumes. The dosimetric parameters collected over the treatment period will be analyzed using linear mixed models with appropriate intra-correlation structures.
Dosimetric changes in lung, heart, and esophageal dosimetry parameters in patients treated with adaptive radiation planning | Baseline up to day 29 of treatment
  Will be compared to computed tomography simulation without adaptation of tumor volumes. The dosimetric parameters collected over the treatment period will be analyzed using linear mixed models with appropriate intra-correlation structures.
Change in toxicities, including cardiac and esophageal toxicities | Baseline up to 25 months after chemoradiation
  Will be compared to historical controls who have not undergo adaptive re-planning at specified time points using Common Terminology Criteria for Adverse Events version 5.0.
Toxicity correlation to disease-free survival (DFS)/progression-free survival (PFS)/overall survival (OS) | Up to 25 months after chemoradiation
  Will determine if toxicity correlates to DFS/PFS/OS using historical controls for comparison, estimated via Kaplan-Meier product limit and compared among different toxicity levels using a log-rank test.
Tumor volume reduction | Up to 25 months after chemoradiation
  Will determine if tumor volume reduction correlates to immunotherapy response.

CONTACTS AND LOCATIONS:
Overall Officials: Salma K Jabbour, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No